CLINICAL TRIAL: NCT00932438
Title: Drug-Eluting Bead, Irinotecan (DEBIRI) Therapy of Liver Metastasis From Colon Cancer With Concomitant Systemic Oxaliplatin, Fluorouracil and Leucovorin Chemotherapy, and Anti-Angiogenic Therapy
Brief Title: Drug-Eluting Bead, Irinotecan (DEBIRI) Therapy of Liver Metastasis From Colon Cancer With Systemic Fluorouracil, Oxaliplatin, Leucovorin and Bevacizumab
Acronym: DEBIRI
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Louisville (Other)
Collaborators: Biocompatibles UK Ltd (Industry)
Responsible Party: Principal Investigator, Robert C. Martin, Professor, University of Louisville
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DEBIRI # 09.0034; UL2008.1
Record Dates: First submitted 2009-07-01; First posted 2009-07-03 (Estimated); Results first posted 2021-05-07 (Actual); Last update posted 2021-06-11 (Actual); Status verified 2018-03

CONDITIONS: Colon Cancer With Metastases to the Liver
Keywords: colon cancer; liver metastases
MeSH Terms: conditions — Colonic Neoplasms | interventions — Oxaliplatin; Folfox protocol; Leucovorin; Fluorouracil; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LC Beads loaded with Irinotecan and FOLFOX6 (Experimental): Device: LC Beads loaded with 100mg Irinotecan
  Drug: Systemic Chemotherapy (FOLFOX6) Oxaliplatin 85 mg/sqm, IV infusion every two weeks Leucovorin 200mg/sqm, IV infusion every two weeks 5-Fluorouracil 2400mg/sqm, IV infusion every two weeks Bevacizumab 5mg/kg given at the discretion of treating physician
  Interventions: Device: LC beads loaded with Irinotecan; Drug: Oxaliplatin; Drug: Leucovorin; Drug: 5-Fluorouracil; Drug: Bevacizumab
- FOLFOX6 and Bevacizumab (Active Comparator): Drug: Systemic Chemotherapy (FOLFOX6) Oxaliplatin 85 mg/sqm, IV infusion every two weeks Leucovorin 200mg/sqm, IV infusion every two weeks 5-Fluorouracil 2400mg/sqm, IV infusion every two weeks Bevacizumab 5mg/kg given at the discretion of treating physician
  Interventions: Drug: Oxaliplatin; Drug: Leucovorin; Drug: 5-Fluorouracil; Drug: Bevacizumab

INTERVENTIONS:
Device: LC beads loaded with Irinotecan — Chemoembolization using LC beads loaded with 100mg Irinotecan
  Other Names: LC Beads, TACE
  Arms: LC Beads loaded with Irinotecan and FOLFOX6
Drug: Oxaliplatin — Oxaliplatin 85 mg/sqm, IV infusion every two weeks
  Other Names: FOLFOX6
Drug: Leucovorin — Leucovorin 200 mg/sqm, IV infusion every two weeks
  Other Names: FOLFOX6
Drug: 5-Fluorouracil — 5-Fluorouracil 2400 mg/sqm, IV infusion every 2 week
  Other Names: FOLFOX6
Drug: Bevacizumab — Bevacizumab 5 mg/kg given at the discretion of the treating physician
  Other Names: Avastin

SUMMARY:
This is a multicentre, open labeled, controlled phase study designed to assess effectiveness of chemoembolization with LC Beads, both with and without systemic chemotherapy, in the treatment of unresectable liver metastases in patients with colorectal cancer.

DETAILED DESCRIPTION:
This is a multicentre, open labeled, prospective, randomized, controlled phase I/II study designed to assess the clinical performance of chemoembolization with Low Compression Bead (LC Bead), loaded with irinotecan in combination with intravenous chemotherapy and bevacizumab versus intravenous chemotherapy in combination with bevacizumab in the treatment of unresectable liver metastases in patients with colorectal cancer.

ELIGIBILITY:
Inclusion:

* Patients over 18 years of age, of any race or sex, who have histologic or radiologic proof of colorectal cancer to the liver, who are able to give informed consent, will be eligible.
* Patients with at least one measurable liver metastases, with size > 1cm response evaluation criteria in solid tumors (RECIST)
* Patients with liver dominant disease defined as ≥80% tumor body burden confined to the liver
* Patients with patent main portal vein
* Eastern Cooperative Oncology Group (ECOG) Performance Status score of < 2
* Life expectancy of > 3 months
* Non-pregnant with an acceptable contraception in premenopausal women.
* Hematologic function: absolute neutrophil count (ANC) ≥ 1.5 x 109/L, platelets ≥75 x109/L, international normalized ratio (INR) ≤1.3* (*If patient is on anticoagulants, they must be able to stop medication temporarily prior to TACE and must have INR ≤1.3 prior to receiving TACE) Adequate liver function as measured by: Total bilirubin ≤ 2.0mg/dl, alanine aminotransferase (ALT), aspartate aminotransferase (AST) ≤5 times upper limits of normal (ULN), albumin ≥2.5g/dl, Adequate Hemoglobin and Hematocrit as measured by (Male: for approximate 45 - 62%; and approximate Female: 37 - 48%) or Hemoglobin (Male: approximate 13 - 18 gm/dL Female: approximate 12 - 16 gm/dL). If patient is asymptomatic with Hemoglobin for male 10 to 12.9 or Female 9.5 to 11.9 and do not wish to be transfused they still will be eligible for treatment.
* Adequate renal function (creatinine ≤ 2.0mg/dl)
* Women of child bearing potential and fertile men are required to use effective contraception negative serum beta human chorionic gonadotropin (βHCG)
* Signed, written informed consent
* Patient is at least one month out from any treatment for Stage III colorectal cancer
* Patient is at least one year out from any treatment for their Stage IV colorectal cancer.

  - these patients should not be candidates for curative treatments, and will have recovered from any chemotherapeutic toxicities' they may have experienced."
* Less than 60% liver tumor replacement

Exclusion:

* "Any patient eligible for curative treatment (i.e. resection or radiofrequency ablation). Note: resectability is defined as a single tumor <5cm with adequate liver function defined: Total bilirubin ≤ 2.0mg/dl" non-resectability includes patients with greater than 6, tumors close to blood vessels, patients with hepatic-pulmonary shunting, or patients of poor performance"
* Active bacterial, viral or fungal infection within 72 hours of study entry
* Women who are pregnant or breast feeding
* Allergy to contrast media that cannot be managed with standard care (e.g. steroids), making magnetic resonance imaging (MRI) or computed tomography (CT) contraindicated.
* Presence of another malignancy with the exception of cervical carcinoma in situ and stage I basal or squamous carcinoma of the skin.
* Any contraindication for hepatic embolization procedures:

  * Large shunt as determined by the investigator (pretesting with TcMMA not required)
  * Severe atheromatosis
  * Hepatofugal blood flow
  * Main portal vein occlusion (e.g. thrombus or tumor)
* Other significant medical or surgical condition, or any medication or treatment, that would place the patient at undue risk and that would preclude the safe use of chemoembolization or would interfere with study participation
* Patients with prior contraindications for the use of irinotecan therapy-this would include chronic inflammatory bowel disease and or bowel obstruction, history of severe hypersensitivity reactions to irinotecan hydrochloride, trihydrate, lactic acid or to any of the excipients of camptosar, severe bone marrow failure, history of Gilbert Syndrome or concomitant use with St. John's Wort
* Patients with prior contraindications for the use of fluorouracil, oxaliplatin, leucovorin or bevacizumab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2009-06; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert CG Martin, MD, PhD, Study Director — University of Louisville
Locations (10):
- United States (9):
  - Clearview Cancer Center, Huntsville, Alabama
  - Radiology Associates of Sacramento/Sutter Cancer Center, Sacramento, California
  - Emory University, Atlanta, Georgia
  - Northside Hospital/GA Cancer Specialists, Atlanta, Georgia
  - University of Louisville, Louisville, Kentucky
  - Hematology and Oncology Assoc. at Bridgeport, Tupelo, Mississippi
  - Washington University/Alvin J. Siteman Cancer Center, St Louis, Missouri
  - Providence Portland Medical Center/Providence Cancer Center, Portland, Oregon
  - Froedtert Memorial Lutheran Hospital, Milwaukee, Wisconsin
- Hospital Italiano de Buenos Aires, Buenos Aires, Argentina

RESULTS

PARTICIPANT FLOW:
Groups:
- Irinotecan Beads With FOLFOX6: LC bead loaded with Irinotecan: Chemoembolization using LC beads loaded with 100mg Irinotecan in combination with Fluorouracil, Oxaliplatin, Leucovorin and Avastin alternating on a 2 week schedule
- FOLFOX6/Avastin Alone: FOLFOX6 and Avastin: Fluorouracil, Oxaliplatin, Leucovorin and Avastin given biweekly
Period: Overall Study
Arm/Group | Irinotecan Beads With FOLFOX6 | FOLFOX6/Avastin Alone
Started | 40 | 30
Completed | 39 | 30
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- LC Beads Loaded With Irinotecan and FOLFOX6: Device: LC Beads loaded with 100mg Irinotecan
  Drug: Systemic Chemotherapy (FOLFOX6) Oxaliplatin 85 mg/sqm, IV infusion every two weeks Leucovorin 200mg/sqm, IV infusion every two weeks 5-Fluorouracil 2400mg/sqm, IV infusion every two weeks Bevacizumab 5mg/kg given at the discretion of treating physician
  LC bead loaded with Irinotecan: Chemoembolization using LC beads loaded with 100mg Irinotecan
  Oxaliplatin
  Leucovorin
  5-Fluorouracil
  Bevacizumab
- FOLFOX6 and Bevacizumab: Drug: Systemic Chemotherapy (FOLFOX6) Oxaliplatin 85 mg/sqm, IV infusion every two weeks Leucovorin 200mg/sqm, IV infusion every two weeks 5-Fluorouracil 2400mg/sqm, IV infusion every two weeks Bevacizumab 5mg/kg given at the discretion of treating physician
  Oxaliplatin
  Leucovorin
  5-Fluorouracil
  Bevacizumab
- Total: Total of all reporting groups
Arm/Group | LC Beads Loaded With Irinotecan and FOLFOX6 | FOLFOX6 and Bevacizumab | Total
Number analyzed (Participants) | 40 | 30 | 70
Age, Continuous [Median (Full Range); unit: years] | 57 [18 to 80] | 60 [18 to 80] | 58.5 [18 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 21 | 37
  Male | 24 | 9 | 33
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 4 | 11
  White | 33 | 25 | 58
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Argentina | 1 | 0 | 1
  United States | 39 | 30 | 69

OUTCOME MEASURES:

1. Primary Outcome: Tumor Response
Description: Tumor response will be determined using Modified Response Evaluation Criteria in Solid Tumors (mRECIST). Response will classified as: Complete response - disappearance of all lesions; Partial response - at least 30% decrease in the sum of the longest diameter of target lesions, taking as reference the baseline sum of longest diameter or 30% reduction of arterial enhancement; Progressive disease - at least 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest longest diameter recorded since start of treatment or appearance of one or more new lesions greater than 1cm in size; Stable disease - neither sufficient shrinkage to qualify for partial response nor sufficient increase to qualify for progressive disease, taking as reference the smallest sum longest diameter since start of treatment.
Time Frame: Months 2, 4 and 6
Population: Intent to treat population: all randomized subjects who received at least one cycle of intravenous chemotherapy or LC bead loaded with irinotecan
Measure: Number; unit: participants
Arm/Group | LC Beads Loaded With Irinotecan and FOLFOX6 | FOLFOX6 and Bevacizumab
Number analyzed (Participants) | 40 | 30
participants | 31 | 16

2. Secondary Outcome: Number of Serious Adverse Events
Description: Total number of serious adverse events that occurred in both Arms of the study.
Time Frame: First treatment through one year post treatment completion
Population: Any subject who received at least one bead treatment in Arm 1 and any subject who received at least one dose of chemotherapy in Arm 2
Measure: Number; unit: Serious Adverse Event
Arm/Group | Irinotecan Beads With FOLFOX6 | FOLFOX6/Avastin Alone
Number analyzed (Participants) | 40 | 30
Serious Adverse Event | 49 | 21

ADVERSE EVENTS:
Arm/Group | LC Beads Loaded With Irinotecan and FOLFOX6 | FOLFOX6 and Bevacizumab
All-Cause Mortality (participants affected / at risk) | 30/40 | 18/30
Serious Adverse Events (participants affected / at risk) | 40/40 | 20/30
Other Adverse Events (participants affected / at risk) | 40/40 | 30/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | LC Beads Loaded With Irinotecan and FOLFOX6 (N=40) | FOLFOX6 and Bevacizumab (N=30)
GU Obstruction (Renal and urinary disorders) | 2 (2) | 2 (2)
PRES Syndrome (Vascular disorders) | 3 (3) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2)
Bowel Obstruction (Gastrointestinal disorders) | 3 (3) | 1 (1)
Renal Failure (Renal and urinary disorders) | 4 (4) | 3 (3)
Necrotizing Cholecystitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 7 (7) | 6 (6)
Hypertension (Vascular disorders) | 4 (4) | 1 (1)
Allergic Reaction (Immune system disorders) | 2 (2) | 0 (0)
Colonic Portal Obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hypokalemia (General disorders) | 1 (1) | 0 (0)
Confusion (General disorders) | 1 (1) | 0 (0)
Bowel Perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dehydration (General disorders) | 6 (6) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 2/30 (2) | 0 (0)
Sepsis (Infections and infestations) | 3 (3) | 0 (0)
Viral Respiratory Infection (Infections and infestations) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pain Back (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Thrombus (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Fever (General disorders) | 1 (1) | 0 (0)
Small Bowel Fistula (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pulmonary Emboli (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Colostomy Perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Cholecystitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Chest Pain (Cardiac disorders) | 1 (1) | 0 (0)
Groin Hematoma (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Weakness (General disorders) | 2 (2) | 0 (0)
Hypokalemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LC Beads Loaded With Irinotecan and FOLFOX6 (N=40) | FOLFOX6 and Bevacizumab (N=30)
Anemia (Blood and lymphatic system disorders) | 12 (12) | 4 (4)
Diarrhea (Gastrointestinal disorders) | 9 (9) | 6 (6)
Vomiting (Gastrointestinal disorders) | 4 (4) | 4 (4)
Nausea (Gastrointestinal disorders) | 9 (9) | 4 (4)
abdominal Pain (Gastrointestinal disorders) | 9 (9) | 3 (3)
Constipation (Gastrointestinal disorders) | 6 (6) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 4 (4) | 2 (2)
Gastritis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (2) | 5 (5)
Depression (Psychiatric disorders) | 2 (2) | 1 (1)
Anxiety (Psychiatric disorders) | 4 (4) | 0 (0)
Altered Mental Status (Psychiatric disorders) | 4 (4) | 0 (0)
Allergic Reaction (Immune system disorders) | 1 (1) | 3 (3)
Herpes Zoster (Immune system disorders) | 3 (3) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 4 (4) | 5 (5)
Tachycardia (Cardiac disorders) | 4 (4) | 2 (2)
Arrythmia (Cardiac disorders) | 2 (2) | 0 (0)
Hypertension (Vascular disorders) | 8 (8) | 6 (6)
Increased Blood Pressure (Vascular disorders) | 11 (11) | 2 (2)
Pulmonary Emboli (Vascular disorders) | 1 (1) | 2 (2)
Somnolence (Psychiatric disorders) | 2 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Fatigue (General disorders) | 16 (16) | 15 (15)
Decreased Appetite (General disorders) | 2 (2) | 0 (0)
Weight Loss (General disorders) | 4 (4) | 1 (1)
Chest Pain (General disorders) | 3 (3) | 0 (0)
Chills (General disorders) | 3 (3) | 1 (1)
Edema (General disorders) | 2 (2) | 2 (2)
Thrombocytopenia (Investigations) | 7 (7) | 2 (2)
Hypokalemia (Investigations) | 4 (4) | 3 (3)
Neutropenia (Investigations) | 6 (6) | 7 (7)
Hyperbilirubinemia (Investigations) | 2 (2) | 1 (1)
Hyponatremia (Investigations) | 3 (3) | 0 (0)
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 9 (9)
Dysphagia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Stomatitis (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 5 (5)
Rash (Skin and subcutaneous tissue disorders) | 9 (9) | 6 (6)
Alopecia (Skin and subcutaneous tissue disorders) | 9 (9) | 4 (4)
Pruritis (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (3)
Diaphoresis (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Dry Skin (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 9 (9) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 6 (6) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 5 (5)
Headache (Nervous system disorders) | 4 (4) | 2 (2)
Neuropathy (Metabolism and nutrition disorders) | 16 (16) | 23 (23)
Dizziness (Nervous system disorders) | 2 (2) | 3 (3)
Parasthesia (Nervous system disorders) | 4 (4) | 4 (4)
Urinary Retention (Renal and urinary disorders) | 0 (0) | 2 (2)
Dysuria (Renal and urinary disorders) | 2 (2) | 0 (0)
Ascites (Hepatobiliary disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No